CLINICAL TRIAL: NCT04191590
Title: Impact of Chronic Rhinosinusitis on the Index of Ciliary Beat Efficiency Using Fluorescent Nanosticks
Brief Title: Impact of Chronic Rhinosinusitis on the Index of Ciliary Beat Efficiency Using Fluorescent Nanosticks: (R-IMPAC)
Acronym: R-IMPAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid crisis
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Foundation for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R-IMPAC
Record Dates: First submitted 2019-12-05; First posted 2019-12-10 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with Chronic Rhinosinusitis (CRS) (Other): Patients with endonasal surgery scheduled under general anesthesia for an indication of Chronic Rhinosinusitis (CRS)
  Interventions: Procedure: nasal brushing and bacteriological sample
- Patient without Chronic Rhinosinusitis (CRS) (Other): Patients with endonasal surgery scheduled under general anesthesia for an indication of endonasal surgery for nasal obstruction or patients requiring an endonasal surgical approach such as pituitary adenomas for example.
  Interventions: Procedure: nasal brushing and bacteriological sample

INTERVENTIONS:
Procedure: nasal brushing and bacteriological sample — A nasal brushing as well as a bacteriological sample using a swab under general anesthesia at the beginning of the endonasal surgery procedure

SUMMARY:
Impact of chronic rhinosinusitis on the index of ciliary beat efficiency using fluorescent nanosticks

DETAILED DESCRIPTION:
To date, the assessment of ciliary beat is only possible ex vivo on epithelial cells obtained from upper airway brushing. A previous prospective study (I-IsBac) showed a change in ciliary beat (in terms of coordination and frequency) in bacterial rhinosinusitis. The study of ex-vivo ciliary movement appears to be an interesting tool to understand the pathophysiology of CSRs and to guide and evaluate treatment.

A new tool to evaluate the effectiveness of the ex-vivo lash beat has been developed. This tool measures shear stress by tracking balls along the ciliary margin.

This measurement of ex-vivo shear stress by bead tracking is a validated technique. However, microbead tracking is limited by its low spatial and temporal resolution, long measurement time and heavy post-processing of acquisition data, making this method difficult to use in clinical routine. Monitoring ex-vivo fluorescent nano-batons could represent a simpler alternative for the clinician. This measurement is now made possible by Phosphate Lanthanum Lanthanum Nano-batons (LaPO4) whose luminescence is directly proportional to the shear.

The objective of this research project is to validate this new tool in patients with CSR by comparing it to a group of control subjects free of nasal inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥ 18 years old

   * Having chronic rhinosinusitis (RCS) requiring surgical treatment. Or
   * With an indication for endonasal surgery for nasal obstruction (turbinoplasty and septoplasty) or for an endonasal surgical approach
2. Acceptance to participate in the protocol with signed informed consent
3. Affiliated or beneficiary of a social security scheme

Exclusion Criteria:

1. Refusal to participate in the study
2. No one who does not speak or understand French
3. Pregnant or breastfeeding woman
4. Persons who are incapable of reaching the age of majority, under guardianship, guardianship or protection of justice.
5. Simulated participation in another intervention research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
The shear stresss by tracking nano-batons (mPa) | Day of the surgical procedure under General Anesthesia
  The value of the shear stress by tracking nano-batons in mPa

SECONDARY OUTCOMES:
Mucosal inflammation score (0 to 10) | Inclusion Visit
  Mucosal inflammation score and presence of polyps during endoscopy
Presence of pus at endoscopy | Inclusion Visit
  Presence of pus at endoscopy
Frequency of ciliary beat | Day of the surgical procedure under General Anesthesia
  Frequency of the ciliary beat
Shear stress by Tracking microbeads (mPa) | Day of the surgical procedure under General Anesthesia
  Value of shear stress by tracking microbeads in mPa
Presence of polyps at endoscopy | Inclusion Visit
  Presence of polyps at endoscopy
coordination of cillary beat | Day of the surgical procedure under General Anesthesia
  Cillary beat coordination evaluated by microscopy

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Hôpital Bicêtre, Le Kremlin-Bicêtre

IPD SHARING:
Plan to Share IPD: No